CLINICAL TRIAL: NCT05669807
Title: A Randomized, Controlled, Multicenter Phase II Study of Camrelizumab Combined With Irinotecan or Albumin Paclitaxel for Second-line Treatment of Advanced Gastric Cancer
Brief Title: Camrelizumab Combined With Irinotecan or Albumin Paclitaxel for Second-line Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, MD, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG-2101
Record Dates: First submitted 2022-11-28; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Second Line Treatment of Gastric Cancer
MeSH Terms: interventions — camrelizumab; Albumin-Bound Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Camrelizumab+Albumin-bound paclitaxel (Experimental): Camrelizumab 200mg d1, one cycle every 14 days on the first day; albumin binding paclitaxel: 100 mg/m2, one cycle every 28 days on the first, eighth and fifteenth days
  Interventions: Drug: Camrelizumab; Drug: Albumin-Bound Paclitaxel
- B: Camrelizumab+Irinotecan (Experimental): Camrelizumab 200mg d1, the first day, every 14 days as a cycle Irinotecan: 180 mg/m2, the first day, every 14 days as a cycle
  Interventions: Drug: Camrelizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Camrelizumab — 200mg d1, the first day, every 14 days as a cycle
  Other Names: Camrel
Drug: Albumin-Bound Paclitaxel — 100 mg/m2, the 1st, 8th and 15th days, every 28 days as a cycle
  Other Names: ABP
  Arms: A: Camrelizumab+Albumin-bound paclitaxel
Drug: Irinotecan — 180 mg/m2, the first day, every 14 days as a cycle
  Other Names: Iri
  Arms: B: Camrelizumab+Irinotecan

SUMMARY:
This study is a multicenter, open, and randomized clinical phase II exploratory study. The "pick the winner" study design is used to determine and select which chemotherapy drug (irinotecan vs. albumin plus paclitaxel) is more effective in the second-line treatment of advanced gastric cancer, and it is more hopeful to carry out the follow-up phase III study in the second-line treatment of advanced gastric cancer (karelizumab+chemotherapy vs. chemotherapy). The study plans to include 184 patients with advanced gastric cancer who have received first-line platinum+fluorouracil progression, randomly use albumin paclitaxel+carrelizumab or irinotecan+carrelizumab second-line therapy, and observe the objective effective rate (ORR), total survival time (OS), progression free survival time (PFS), treatment related adverse reactions, quality of life and other clinical indicators after receiving the above treatment, Then determine the second line scheme which is more advantageous.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75
* ECOG score: 0 or 1
* Unresectable advanced or recurrent gastric cancer/gastroesophageal junction cancer
* histologically proven adenocarcinoma
* Received chemotherapy based on platinum and fluorouracil within 12 months
* Patients not previously treated with paclitaxel or irinotecan
* Liver function: total bilirubin, ALT and AST<1.5 × ULN (Normal Value upper limit)
* Renal function: Cr<1.5 × ULN and creatinine clearance ≥ 40 ml/min
* Echocardiography or radionuclide cardiac function test, LVEF ≥ 50%
* Expected survival ≥ 3 months
* Sign the informed consent form

Exclusion Criteria:

* Patients who have received irinotecan or paclitaxel chemotherapy in the past
* ECOG PS score:>2
* Advanced gastric cancer patients with extensive and severe peritoneal metastasis
* Patients with severe liver and kidney insufficiency or cardiac insufficiency
* HIV positive, active hepatitis B or C, active pulmonary tuberculosis
* Patients with active autoimmune diseases, including lupus erythematosus, rheumatoid arthritis, rheumatoid arthritis, etc
* Patients known to be allergic to any of the study drugs
* Pregnant or lactating female patients

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 12 weeks
  CR+PR

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of date of death from any cause, assessed up to 24 months
  Time from random start of treatment to death from any cause
Progression-free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from random start of treatment to death or tumor progression due to any reason
Treatment related adverse reactions | 24 months
  Evaluation according to CTC 4.0
Quality of life assessment | 24 months
  according to EORTC C30

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, Principal Investigator — Zhejiang Cancer Hospital

IPD SHARING:
Plan to Share IPD: No